CLINICAL TRIAL: NCT04186923
Title: Familien-SCOUT: Comprehensive Support for Families With a Parent Suffering From Cancer
Acronym: F-SCOUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-033
Record Dates: First submitted 2019-12-02; First posted 2019-12-05 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Families With Minor Children and One Parent Suffering From Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (IG) (Experimental): Families receive permanent contact persons to support in the organisation of everyday life, financial applications, during emotional coping with illness and open communication within the family.
  Interventions: Other: F-SPOKE
- Control Group (No Intervention): In the control group the families are treated according to the standard of care.

INTERVENTIONS:
Other: F-SPOKE — This project includes communicative, emotional, and also organizational support with outreach across different sectors and phases (F-SPOKE - family-centered, cross-sector and cross-phase organizational, communicative, and emotional support).
  Arms: Intervention group (IG)

SUMMARY:
When a parent with minor children falls ill with cancer, it is extremely stressful for all of the family members, including the partner and children. Familiar everyday routines are often disrupted even at an early stage, and for a prolonged period. Financial difficulties, the threat represented by the uncertain course of the disease, and worries about the children's future have a cumulative effect. The affected families are thereby pushed to their limits organizationally and emotionally. The burden involved tends to be underestimated, and secondary psychological conditions often develop among all the family members. They often do not have adequate access to support.

The aim of this project is to establish a care management system that provides support for families with underage children in which one parent is seriously ill. In order to reduce the burden on families, "family SCOUTS" are to be used who can provide advice and information at an early stage. They are intended to encourage families to discuss things openly, and they should also facilitate access to all the support services available.

The project will evaluate whether the use of family SCOUTS reduces the burden on the family in comparison with families who do not have a family SCOUT. For this purpose, investigations will be carried out before and after the family SCOUTS are deployed. Standardized questionnaires, interviews, and routine data from the participating health-insurance companies will provide the basic data.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed ICD diagnosis of cancer in one parent
* Custody of at least one underage child
* Adequate knowledge of German
* Availability of informed consent to participate in the study from the patient and/or healthy parent and linkage to questionnaire data and routine data

Exclusion Criteria:

* Withdrawal of consent by the ill or healthy parent
* Relevant cognitive limitation, advanced dementia
* Individuals who are in relationships of dependence or employment to the project managers or their representatives

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS | Change from Baseline HADS at 9 months
  HADS is used to record anxiety and depression in patients with physical diseases or psychogenic physical symptoms.Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. The HADS uses a scale and therefore the data returned from the HADS is ordinal.

SECONDARY OUTCOMES:
Distress Thermometer (DT) | baseline & 9 month
  DT is a screening instrument developed by the National Comprehensive Cancer Network (NCCN) for registering psychosocial stress in oncological patients. It consists of a scale from 0 to 10 and a list of problems, providing a scheme for referral to the relevant professional services.
Parenting Concerns Questionnaire (PCQ) | baseline and 9 month
  PCQ is used to record concerns among parents who have developed cancer. It includes 15 items with a 5-level response scale.
HLS-EU-Q16 | 3 month
  HLS-EU-Q16 measures health competenceliteracy, using 16 items and a four-level response scale.
PA-F-P-KF | baseline & 9 month
  The short form of the Fear of Progression Anxiety Questionnaire for Partners (PA-F-P-KF) records anxieties regarding progression fear of progression in healthy partners of individuals with chronic disease. The scale includes 12 items, each with a 5-level scale of response categories.
CaPIN | 3 & 9 Month
  The Cancer Patient Information Needs (CaPIN) scale measures information needs on various topics among cancer patients. The scale consists of 22 items with binary-coded response categories (yes/no).
MOS-SS | 3 month
  This instrument is a subscale of the validated "Medical Outcomes Study Social Support (MOS-SS) survey. The eight items on the subscale record emotional and informational social support. The response categories have a five-level scale.
FAD | baseline & 9 month
  The Family Assessment Device (FAD)is based on the McMaster Model of Family Functioning (MMFF), a clinically oriented conceptualization of families. It is a screening instrument only consisting of 53-items. The model identifies six dimensions of family functioning. Scores range from 1 to 4 with 1 reflecting healthy functioning and 4 reflecting unhealthy functioning. The FAD is made up of seven scales.
EQ-5D-5L | baseline, 3 & 9 month
  The EuroQoL Group (EQ)-5D is a generic measurement instrument that uses a standardized, preference-based procedure to describe and investigate health-related quality of life.The EQ-5D-5L is composed of the EQ-5D-5L descriptive system and the EQ Visual Analogue scale (EQ VAS). The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Each level corresponds to 1-digit number expressing the level selected for that dimension.
KIDSCREEN-10: | baseline & 9 month
  The KIDSCREEN questionnaire for children is used to record health-related quality of life (HRQoL). The scale ranges from 5 to 50, with a higher score indicating a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Tim H. Brümmendorf, Prof. Dr., Principal Investigator — Department of Hematology, Oncology, Hemostaseology, RWTH Aachen University
Locations (3):
- Germany (3):
  - Department of Hematology, Oncology, Hemostaseology and Stem Cell Transplantation, Faculty of Medicine, RWTH Aachen University, Aachen
  - Department of Psychosomatic Medicine and Psychotherapy, University Hospital Bonn, Bonn
  - Clinical Institute of Psychosomatic Medicine and Psychotherapy, Heinrich-Heine-University Duesseldorf, Düsseldorf

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holsteg S, Klett MK, Kisic AM, Horbach-Bremen R, Brune M, Dohmen M, Drueke B, Ernstmann N, Geiser F, Heier L, Heuser C, Icks A, Panse J, Petermann-Meyer A, Viehmann A, Karger A. Psychological burden, quality of life, problems, and parental concerns of single mothers with cancer: a cross-sectional comparison. Support Care Cancer. 2025 Feb 11;33(3):173. doi: 10.1007/s00520-025-09225-y. PMID 39932595
- [Derived] Ernstmann N, Nakata H, Heier L, Heuser C, Dohmen M, Bremen R, Geiser F, Holsteg S, Karger A, Viehmann A, Brune M, Icks A, Haastert B, Brummendorf TH, Petermann-Meyer A. Feasibility of a complex psychosocial intervention for families with parental cancer: acceptability, suitability, implementability, and perceived support. J Cancer Res Clin Oncol. 2024 Oct 17;150(10):464. doi: 10.1007/s00432-024-05946-5. PMID 39414623
- [Derived] Heuser C, Schneider JN, Heier L, Ernstmann N, Nakata H, Petermann-Meyer A, Bremen R, Karger A, Icks A, Brummendorf TH, Geiser F. Family resilience of families with parental cancer and minor children: a qualitative analysis. Front Psychol. 2024 Jan 19;14:1251049. doi: 10.3389/fpsyg.2023.1251049. eCollection 2023. PMID 38314254
- [Derived] Dohmen M, Petermann-Meyer A, Blei D, Bremen R, Brock-Midding E, Brune M, Geiser F, Haastert B, Halbach SM, Heuser C, Holsteg S, Heier L, Icks A, Karger A, Montalbo J, Nakata H, Panse J, Rottmann TP, Sattler K, Viehmann A, Vomhof M, Ernstmann N, Brummendorf TH. Comprehensive support for families with parental cancer (Family-SCOUT), evaluation of a complex intervention: study protocol for a non-randomized controlled trial. Trials. 2021 Sep 15;22(1):622. doi: 10.1186/s13063-021-05577-y. PMID 34526078